CLINICAL TRIAL: NCT00854867
Title: Phase I Randomised Multi-centre Study to Demonstrate the Safety of WBRT Concomitant to Intrathecal Liposomal Cytarabine (DepoCyte®) Versus WBRT & Sequential Intrathecal Liposomal Cytarabine (DepoCyte®) for Treatment of STNM With or Without Brain Metastasis.
Brief Title: Study to Demonstrate the Safety of WBR Administered at the Same Time as Intrathecal Liposomal Cytarabine (DepoCyte®) Versus Intrathecal Liposomal Cytarabine (DepoCyte®) Administered After WBR for the Treatment of Solid Tumour Neoplastic Meningitis in Patients With or Without Brain Metastasis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEP1501; 2008-007206-10
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-02

CONDITIONS: Solid Tumour Neoplastic Meningitis; Brain Metastases
Keywords: Solid tumour neoplastic meningitis; STNM; leptomeningeal metastases; DepoCyte; WBRT; Whole Brain Radiotherapy; Liposomal cytarabine intrathecal; Solid Tumour Neoplastic Meningitis with or without brain metastasis
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole brain radiotherapy (WBRT) with concomitant Depocyte (Experimental): Subjects will receive a total of 38.4 Gray (Gy) WBRT given over 4 weeks. Subjects will receive 3 GyWBRT on Days 1 and 2 and then 1.8 Gy on the third fourth and fifth days of WBRT treatment during Week 1. Subjects will then receive 1.8 Gy WBRT per day; 5 days out of seven, each week for the next 3 weeks. A total of 4 doses of DepoCyte (50 mg of liposomal ARA-C) will be administered intrathecally. The first dose will be administered on Day 3 (or Day 4 or 5) of Week 1, i.e. the third day of radiotherapy treatment when the dosage is reduced to 1.8 Gy. The second dose will be administered on Day 17(+2 days); the third dose will be administered on Day 31 (+2 days); the fourth dose will be administered on Day 45 (+2 days) to complete the induction phase of the protocol. Subjects will continue to receive an additional 6 doses of DepoCyte one dose every 28 days (+2 days) during the maintenance period. The first dose will be given 28 days after the last dose in the induction phase.
  Interventions: Drug: Whole brain radiotherapy (WBRT) with concomitant Depocyte
- Whole Brain Radio Therapy (WBRT) with sequential Depocyte (Active Comparator): Subjects will receive a total of 38.4 Gy WBRT given over 4 weeks. Subjects will receive 3 Gy (WBRT on Day 1 and Day 2) and then 1.8 Gy on the third fourth and fifth days of WBRT treatment during Week 1. Subjects will then receive 1.8 Gy WBRT per day; 5 days out of seven, each week for the next 3 weeks. A total of 4 doses of DepoCyte (50 mg of liposomal ARA-C) will be administered intrathecally. The first dose will be administered on Day 29 (+2 days); the second dose will be administered on Day 43(+2 days); the third dose will be administered on Day 57 (+2 days); the fourth dose will be administered on Day 71 (+2 days) to complete the induction phase of the protocol. DepoCyte should never be administered more frequently than every 14th day. Subjects will continue to receive an additional 6 doses of DepoCyte one dose every 28 days (+2 days) during the maintenance period. The first dose will be given 28 days after the last dose in the induction phase.
  Interventions: Drug: Whole Brain Radio Therapy (WBRT) with sequential Depocyte

INTERVENTIONS:
Drug: Whole Brain Radio Therapy (WBRT) with sequential Depocyte
  Arms: Whole Brain Radio Therapy (WBRT) with sequential Depocyte
Drug: Whole brain radiotherapy (WBRT) with concomitant Depocyte
  Arms: Whole brain radiotherapy (WBRT) with concomitant Depocyte

SUMMARY:
The purpose of this study is to demonstrate the safety of giving Whole Brain Radiotherapy (WBRT) together with intrathecal liposomal cytarabine (DepoCyte®) for patients with leptomeningeal metastases. The study will compare the safety of giving DepoCyte at the same time as WBRT with giving the drug after WBRT is complete.

ELIGIBILITY:
Indication and Criteria for Inclusion/Exclusion:

Subjects who are to be included in the study have to meet all of the following criteria:

* Informed consent
* Male and female, age over 18 years
* Solid tumour neoplastic meningitis as demonstrated by a positive lumbar CSF cytology (obtained within 21 days prior to treatment initiation) OR Characteristic signs and symptoms of neoplastic meningitis PLUS an MRI indicating the presence of meningeal tumour (diagnosis to be made by neuro-oncologist and confirmed / signed within the CRF). All MRIs will be forwarded for central review and confirmation of diagnosis. In case of discrepancy the central review overrides the assessment of the investigator.
* CSF flow abnormality excluded by either an MRI scan or a 99Tc-DTPA or 111In-DTPA flow study.

(If a flow abnormality is initially demonstrated but the flow block is subsequently documented by another flow study or MRI scan to be relieved following limited field radiation therapy, the subject may then be eligible)

* If brain metastasis confirmed (including subjects who have had previous stereotactical radiosurgery or solitary lesion brain surgery) the lesion should be less than 3cm diameter
* Mini Mental State Examination (MMSE) score more than 24
* ECOG performance status 0-2

Laboratory values as follows:

* Platelet count more than or equal to 80,000/mm3
* ANC more than or equal to 1,000/mm3
* Serum creatinine less than or equal to 2 x upper limit of normal
* Total bilirubin less than or equal to 3 x upper limit of normal
* SGOT (AST) less than or equal to 3 x upper limit of normal
* LDH less than or equal to 3 x upper limit of normal

  * Females of child-bearing potential must have a negative (urine or serum) pregnancy test within 21 days prior to the start of study treatment.
  * Females of childbearing potential must be willing to use an effective method of contraception to prevent pregnancy for the duration of the study (e.g. implants, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence or vasectomised partner).
  * Males must be willing to use an effective method of contraception with their partner to prevent pregnancy for the duration of the study (e.g. implants, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence or vasectomy).

Exclusion Criteria:

* Previous WBRT
* Brain metastases more than 3 cm diameter
* Previous IT treatment
* Uncontrolled infection including HIV infection
* Any present condition that is regarded as contraindication for WBRT and intrathecal chemotherapy
* Prior treatment with systemic ARA-C
* Anticipated hypersensitivity to DepoCyte or ARA-C
* Clinically manifest encephalopathy
* On anticoagulant therapy
* Ventricular peritoneal CSF drain in situ
* Subjects unable to comply with study procedures
* Pregnancy and lactation Any other investigational drug administered within 21 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate that WBRT concomitant to DepoCyte is as safe as WBRT & sequential DepoCyte in treating solid tumour neoplastic meningitis with/without brain metastasis. | Safety is reviewed at every visit & for 3 months after last Depocyte administration

SECONDARY OUTCOMES:
Overall response rate (ORR) | Safety is reviewed at every visit & for 3 months after last Depocyte administration
Progression free survival (PFS) | Safety is reviewed at every visit & for 3 months after last Depocyte administration
Time to neurologial progression (TNP) | Safety is reviewed at every visit & for 3 months after last Depocyte administration
Overall survival (OS) | Safety is reviewed at every visit & for 3 months after last Depocyte administration

CONTACTS AND LOCATIONS:
Locations (7):
- Austria (6):
  - Feldkirch Regional Hospital, Feldkirch
  - Graz Medical University, Graz
  - Univeristy Clinic for Radiotherapy and Radio-Oncology, Innsbruck
  - Klagenfurt Regional Hospital, Klagenfurt
  - University Internal Medicine Clinic III, Salzburg
  - Kaiser-Franz-Josef-Spital, Vienna
- Heidelbert, Germany

REFERENCES:
- See also: Results available on website — http://www.mundipharma-rd.eu